CLINICAL TRIAL: NCT05240352
Title: Developing Brain Imaging Analysis Expertise for Personalizing Transcranial Electric Stimulation in Anhedonia Treatment of Patients with Bipolar Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Milken Institute (Other)
Responsible Party: Principal Investigator, Jair Soares, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-21-1044
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Anhedonia
Keywords: bipolar depression
MeSH Terms: conditions — Anhedonia; Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- active tDCS (Experimental)
  Interventions: Device: active tDCS
- sham tDCS (Sham Comparator)
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: active tDCS — Subjects will receive active dose (constant current intensity of 2mA) from the tDCS device for 30 minutes per session for two weeks with no sessions on Saturday and Sunday (Monday to Friday), and one additional session two and four weeks later
  Arms: active tDCS
Device: sham tDCS — Subjects will receive a dose from a "sham-tDCS"that is, a device which delivers a different pattern of electric current for 30 minutes per session for two weeks with no sessions on Saturday and Sunday (Monday to Friday), and one additional session two and four weeks later
  Arms: sham tDCS

SUMMARY:
The purpose of this study is to investigate whether transcranial direct-current stimulation (tDCS) will engage reward-related brain circuitry, more specifically the uncinate fasciculus (UF) tract, which connects the orbitofrontal cortex (OFC) and nucleus accumbens (NAcc) regions. Also to evaluate whether the changes in the fractional anisotropy (FA) of the UF tract are associated with changes of clinical symptoms of anhedonia and finally to investigate the moderation role of simulated electric fields (EFs) in an association between FA of the UF and symptoms of anhedonia.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Bipolar Disorder and clinically significant anhedonia
* mild symptoms of depression

Exclusion Criteria:

* substance abuse/dependence and any use of drugs (except alcohol or nicotine) in the previous month of the baseline assessment
* participants with personality disorder that would interfere with study participation according to clinical judgment
* previous neurological conditions (epilepsy, traumatic brain injury, stroke, etc)
* any severe, life-threatening non-psychiatric medical condition
* specific contraindications for tDCS (metallic plates in the head)
* Participants identified as acutely suicidal or severely agitated

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
change in the fractional anisotropy of the uncinate fasciculus | baseline, 6 weeks
  Change in the fractional anisotropy of the uncinate fasciculus as assessed by diffusion tensor imaging (DTI)

SECONDARY OUTCOMES:
changes in symptoms of anhedonia as assessed by the Snaith-Hamilton Pleasure Scale modified for clinical administration (SHAPS-C) | baseline, 6 weeks
  This is a 14 item questionnaire and each is scored from 1 to 4 (1 = Lots of pleasure, 4 = No pleasure)
change in symptoms of anticipatory anhedonia as assessed by the Temporal Experience of Pleasure Scale (TEPS) | baseline, 6 weeks
  The TEPS presents 18 items, 10 of them related to the experience of anticipatory pleasure, and the other 8 related to the ability to experience pleasure at the moment. This is scored on a 6-point Likert scale (1 = very false for me to 6 = very true for me).Total scores vary form 18-108 and lower scores mean higher anhedonia
change in symptoms of consummatory anhedonia as assessed by the Temporal Experience of Pleasure Scale (TEPS) | baseline, 6 weeks
  The TEPS presents 18 items, 10 of them related to the experience of anticipatory pleasure, and the other 8 related to the ability to experience pleasure at the moment. This is scored on a 6-point Likert scale (1 = very false for me to 6 = very true for me).Total scores vary form 18-108 and lower scores mean higher anhedonia

CONTACTS AND LOCATIONS:
Overall Officials: Jair C Soares, MD,PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No